CLINICAL TRIAL: NCT01343745
Title: Dose Response Evaluation of CHF 1535 HFA pMDI in Asthmatic Patients Using Lung Function, Adenosine Monophosphate Bronchial Challenge and Fractional Exhaled Nitric Oxide (FENO)
Brief Title: Dose Response AMP Challenge Study With Beclometasone Dipropionate (BDP)/Formoterol Pressurised Metered Dose Inhaler (pMDI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FB/PS/14/169/07; 2007-004345-14 (EudraCT Number)
Record Dates: First submitted 2011-04-21; First posted 2011-04-28 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Mild Persistent Asthma
MeSH Terms: interventions — Foster Home Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo pMDI
  Interventions: Drug: Placebo
- Low dose (Experimental): BDP/formoterol pMDI low dose
  Interventions: Drug: BDP/formoterol
- High dose (Experimental): BDP/Formoterol pMDI high dose
  Interventions: Drug: BDP/formoterol

INTERVENTIONS:
Drug: BDP/formoterol — pressurised metered dose inhaler, BDP + Formoterol 100/6 µg, 4 inhalations bid (total daily dose 800 µg BDP + 48 µg formoterol)
  Other Names: Foster
  Arms: High dose
Drug: BDP/formoterol — pressurised metered dose inhaler, BDP + Formoterol 100/6 µg, 1 inhalation bid (total daily dose 200 µg BDP + 12 µg formoterol)
  Other Names: Foster
  Arms: Low dose
Drug: Placebo — pressurised metered dose inhaler
  Arms: Placebo

SUMMARY:
The aim of this exploratory investigation is to evaluate if the Forced Expiratory Volume in the 1st second (FEV1) measurements, fractional exhaled nitric oxide (FENO) and Provocative Concentration 20 (PC20) after Adenosine Monophosphate (AMP) bronchial challenge evaluated after administration of a fixed combination of a Long-acting Beta-2-agonist (LABA) and an Inhaled Corticosteroid (ICS) at increasing doses may be suitable to demonstrate a dose response.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18-50 years of age, who have signed an informed consent form.
2. Clinical evidence of asthma
3. Steroid naïve asthmatic patients
4. FEV1 at Screening Visit is >70 % of the predicted value and at least 2.0 L.
5. Body Mass Index between 18 and 35.
6. Sensitivity to AMP at Screening Visit.
7. FENO levels >25 ppb at the Screening Visit

Exclusion Criteria:

1. Having received an investigational product within 2 months of Screening Visit.
2. Inability to comply with study procedures or with study treatment intake.
3. Any significant lung disease which is considered by the investigator to be clinically significant.
4. Patients who suffer from Chronic Obstructive Pulmonary Disease (COPD)
5. Previous or current smokers who have a smoking history greater than 5 pack years.
6. Patients with any uncontrolled disease that might, in the judgment of the investigator, place the patients at undue risk or potentially compromise the results or interpretation of the study.
7. Patients with QTc >450msec at the Screening Visit.
8. Patients with serum potassium <3.5 mEq/L or >6 mEq/L.
9. Intolerance/hypersensitivity or any contra-indication to treatment with beta2-agonists and/or inhaled corticosteroids.
10. Patients who have a history of alcohol or substance abuse that in the opinion of the Investigator may be of clinical significance.
11. Patients who have undergone major surgery in the previous 3 months.
12. Patients who have had an exacerbation of asthma, requiring treatment with oral steroids during the last month prior to Screening Visit.
13. Patients treated with slow-release corticosteroids 2 months prior to Screening Visit.
14. Patients currently treated with anti-IgE Antibodies.
15. Patients who have had a respiratory tract infection within 4-weeks prior to Screening Visit.
16. Females not willing to use effective contraceptive measures such as oral contraceptive or intra-uterine device (IUD).
17. Females who are pregnant, lactating or planning to become pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
PC20 after AMP challenge | 4 h post dose
  Provocative Concentration of AMP causing a 20% fall in FEV1.
Fractional Exhaled Nitric Oxide (FeNO) | 4 h post dose
  Fractional exhaled nitric oxide (ppb). FeNO is a biomarker measured in a breath test and it is a validated method for measuring the airway inflammation in asthma.
Lung function | from 0 to 4 h post dose
  FEV1 area under the curve from 0 to 4 hour post dose (AUC0-4h)

SECONDARY OUTCOMES:
FENO | 2 h post dose
  Fractional exhaled nitric oxide

CONTACTS AND LOCATIONS:
Overall Officials: Brian J O'Connor, MD, Principal Investigator — Heart Lung Centre
Locations (1):
- Respiratory Clinical Trials - Heart Lung Centre - Queen Anne Street Medical Centre, London, United Kingdom

REFERENCES:
- [Result] O'Connor BJ, Collarini S, Poli G, Brindicci C, Spinola M, Acerbi D, Barnes PJ, Leaker B. Rapid effects of extrafine beclomethasone dipropionate/formoterol fixed combination inhaler on airway inflammation and bronchoconstriction in asthma: a randomised controlled trial. BMC Pulm Med. 2011 Dec 21;11:60. doi: 10.1186/1471-2466-11-60. PMID 22188731
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2007-004345-14/results
- See also: CSR Synopsis available in the CHIESI Clinical Study Register — https://www.chiesi.com/clinic/CSR_Synopsis_FB-PS-14-169-07.pdf